CLINICAL TRIAL: NCT06576167
Title: Project IMPROVE: Implementing Community-Engaged Intervention Research to Increase Rapid SARS-CoV-2 Self-Testing Among Diverse Underserved and Vulnerable Asian Americans
Brief Title: COVID-19 Self-testing IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: RADxUP
Record Dates: First submitted 2024-08-27; First posted 2024-08-28 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: stepped wedge clustered-randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wedge 1 (Experimental): The earliest group to implement the IMPROVE intervention ( in 4-9 study months).
  Interventions: Behavioral: IMPROVE
- Wedge 2 (Experimental): Following the wedge 1 group, the wedge 2 group started the intervention in the study months 7-12.
  Interventions: Behavioral: IMPROVE
- Wedge 3 (Experimental): The wedge 3 group started the intervention in the study months 10-15.
  Interventions: Behavioral: IMPROVE

INTERVENTIONS:
Behavioral: IMPROVE — IMPROVE is a CBHN-led intervention. The study team delivered comprehensive training to CHNs to let them be well-prepared for intervention delivery. CHNs lead an in-person start-up group education session that consists of 4 modules: 1) a 6-minutes video of a health care provider delivering information on COVID-19 to help participants better understand the disease; 2) using educational slides, CHNs discuss the importance of COVID-19 testing and mitigation adherence; 3) CHNs conduct live demonstration of how to use rapid COVID-19 self-test kit correctly and distribute two COVID-19 self-testing kits to each participant. 4) CHNs guide interactive discussions with participants to enable them to reflect and reinforce what they learned. In addition, CHNs will help participants identify their navigation needs in reducing hesitancy of self-testing and mitigation practices. CHNs will also schedule check-in calls with participants.

SUMMARY:
The study aims to engage community partners to implement IMPROVE intervention and promote (COVID-19) rapid testing among vulnerable Asian Americans in the Greater Philadelphia Area and New York City

ELIGIBILITY:
Inclusion Criteria:

* (1) self-identified as Asian from one of the subgroups: Chinese, Korean, Vietnamese, Filipino, or other South Asian Americans,
* (2) aged 18 and above,
* (3) living in the Greater Philadelphia or NYC areas,

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1271 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
the change in the rate of COVID-19 self-testing | baseline, 1-month follow up, and 3-month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No